CLINICAL TRIAL: NCT04470050
Title: A Phase 1b/2 Randomized, Double-Blind, Placebo-Controlled, Ascending-Dose Study of BXCL501 to Treat Symptoms of Acute Opioid Withdrawal in Patients With Opioid Use Disorder Who Are Physically Dependent on Opioids
Brief Title: Dexmedetomidine in the Treatment of Symptoms Of Acute Opioid Withdrawal
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioXcel Therapeutics Inc (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BXCL501-201
Record Dates: First submitted 2020-07-01; First posted 2020-07-14 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Opioid Withdrawal
Keywords: Opioid; Opioid Addiction; Opioid Dependance; Opioid Withdrawal Symptoms; Opioid Withdrawal Syndrome; Morphine Addiction; delta-opioid receptors; Inhibition of nociceptive afferent neurons (PNS System); Reduction of nociceptive transmission; Activation of descending inhibitory pathways (CNS System); Analgesic Opioids; Drug craving; μ-δ-opioid (Mu-Delta) receptor; μ-binding (Mu receptors); afferents within laminae I and II; κ-opioid receptor (KOR); δ-opioid receptor (DOR) agonist; (+)-pentazocine; σ receptor antagonists; Downstream involvement of the σ receptor; Increase phosphorylation in p38 MAPK; IL-10; Activation of IL-12; IL-12 increase in T-cell immune response; pentacyclic 3°amine (alkaloid); stereogenic centers; tetrahydroisoquinoline reticuline; CPY2D6; benzylisoquinoline alkaloid; p38 MAPK-dependent pathway; kappa-opioid receptors; Short Opiate Withdrawal Scale (SOWS)-Gossop; Clinical Opiate Withdrawal Scale (COWS); Agitation and Calmness Evaluation Scale (ACES); Discontinuation of Morphine Maintenance
MeSH Terms: conditions — Opioid-Related Disorders; Morphine Dependence; Psychomotor Agitation | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Phase 1b: The blinded opioid maintenance phase (Days 1 to 5). Doses of morphine during Phase 1b varied at the discretion of the investigator, between 120-150 mg per day, depending on patients abuse history and need for a higher dose to stabilize withdrawal symptoms. In addition to morphine maintenance, all subjects received sublingual placebo films, approximately 12 hours apart, at 8 am and 8 pm (30min) during this period to simulate and thus blind treatment to BXCL501 sublingual films during Days 6 to 12 (Phase 2).
  Phase 2: The randomized BXCL501/placebo phase (both active and placebo administered as sublingual films) occurred on Days 6 to 12, followed by 2 days of BXCL501-placebo sublingual film and morphine-placebo capsule treatment for all remaining subjects on Days 13 and 14 following the dosing timeline as administered in the Phase 1b portion of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phase 1b: morphine maintenance, blinded to BXCL501 sublingual treatment (placebo).
  Phase 2: Randomized, Double-blind, placebo-controlled (4:1, active to placebo ratio, respectively).
  Follow-On portion of Phase 2: Double-blind, placebo-controlled (treatment with morphine-placebo capsules and BXCL501-placebo sublingual films as administered during phase 1b)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1- Dexmedetomidine (30 Micrograms) vs. Placebo (Experimental): Sublingual film containing 30 Micrograms Dexmedetomidine or Placebo Sublingual film
  Interventions: Drug: Dexmedetomidine; Drug: Placebo
- Cohort 2- Dexmedetomidine (60 Micrograms) vs. Placebo (Experimental): Sublingual film containing 60 Micrograms Dexmedetomidine or Placebo Sublingual film
  Interventions: Drug: Dexmedetomidine; Drug: Placebo
- Cohort 3- Dexmedetomidine (90 Micrograms) vs. Placebo (Experimental): Sublingual film containing 90 Micrograms Dexmedetomidine or Placebo Sublingual film
  Interventions: Drug: Dexmedetomidine; Drug: Placebo
- Cohort 4- Dexmedetomidine (120 Micrograms) vs. Placebo (Experimental): Sublingual film containing 120 Micrograms Dexmedetomidine or Placebo Sublingual film
  Interventions: Drug: Dexmedetomidine; Drug: Placebo
- Cohort 5- Dexmedetomidine (180 Micrograms) vs. Placebo (Experimental): Sublingual film containing 180 Micrograms Dexmedetomidine or Placebo Sublingual film
  Interventions: Drug: Dexmedetomidine; Drug: Placebo
- Cohort 6- Dexmedetomidine (240 Micrograms) vs. Placebo (Experimental): Sublingual film containing 240 Micrograms Dexmedetomidine or Placebo Sublingual film
  Interventions: Drug: Dexmedetomidine; Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Sublingual Film of Dexmedetomidine
  Other Names: BXCL501
Drug: Placebo — Sublingual Placebo film
  Other Names: Placebo comparator

SUMMARY:
This Phase 1b/2 inpatient study assessed the safety, pharmacokinetics, and early signs of efficacy of escalating doses of BXCL501 versus placebo following discontinuation of morphine maintenance. The opioid (morphine) maintenance phase (Phase 1b) included Days 1-5; the randomized BXCL501/placebo phase (Phase 2) included Days 6-12. The randomized phase was followed by 2 sequential days, Days 13 and 14, utilizing treatment of BXCL501-placebo sublingual films and morphine-placebo capsules for all subjects who remained in the study.

DETAILED DESCRIPTION:
This Study included two phases, Phase 1b and Phase 2. Phase 1b was the morphine maintenance phase, Days 1 through 5 and Phase 2 was the randomized, double-blind, placebo-controlled, ascending-dose study of BXCL501 sublingual films on Days 6-12 to treat symptoms of acute opioid withdrawal in patients with opioid use disorder who are/were physically dependent on opioids. Day 12 was followed by 2 sequential days (Days 13 and 14) of BXCL501 vs. placebo and morphine vs. placebo treatment for all subjects who remained in the study.

After a 30-day screening period, eligible male and female adult subjects with Opioid Use Disorder (OID) who were physically dependent on opioids and were not seeking treatment for opioid withdrawal symptoms were admitted to an inpatient unit. The opioid maintenance phase of the study (Phase 1b, Days 1-5) began on Day 1 and continued through Day 5. Approximately 225 subjects were enrolled in the Phase 1b study in cohorts (approximately 25 subjects/cohort). All subjects enrolled in the Phase 1b portion of the study received oral morphine capsules. The total dose of morphine during the opioid maintenance phase varied at the discretion of the investigator, ranged between 120 mg and 150 mg per day, depending on patients abuse history and need for higher dose to stabilize withdrawal symptoms. In addition, these subjects received placebo sublingual films approximately 12 hours apart to simulate and thus blind treatment of BXCL501 during Phase 2 of the study (Days 6-12).

Abrupt discontinuation of active morphine began on Day 6 (Phase 2) and subjects were randomized in a 4:1 ratio to receive either BXCL501 sublingual films or placebo sublingual films, respectively. 135 subjects enrolled/rolled over from the Phase 1b portion of the study into the randomized, double-blind, placebo-controlled portion of the study (Phase 2). Subjects were treated according to their assigned, randomized treatment from Day 6 through Day 12. Treatment was administered approximately 12 hours apart at approximately 8am (±30 minutes) and 8pm (±30 minutes); the 2nd dose (evening dose) was administered only to subjects that were hemodynamically stable, not hypotensive (must be greater than 110/70 diastolic/systolic), and not bradycardic (must be greater than 55 beats per minute (bpm)). Subjects were not given the second dose if they were orthostatic (a drop of 20 points in either systolic blood pressure (SBP) or 10 points in Diastolic Blood Pressure (DBP)) or if they were experiencing an Adverse Event (AE) that when assessed by the Investigator. If a subject experienced SBP <90 mmHg; or DBT <60 millimeters of mercury (mmHg); or Heart Rate (HR) <50 bpm, immediately prior to the next dose, administration of the study medication for that subject was withheld until resolution of the BP and HR parameters. The administration hold did not exceed 2 hours. Safety and tolerability were monitored continuously and summarized upon completion of each cohort by medical safety review.

Studies of opioid withdrawal with placebo arms are likely to have high dropout rates, thus, the dropouts prior to Day 6 could be replaced to ensure enough sample size entering the treatment phase in Phase 2. Dropouts after Day 6 were not to be replaced. The study was intended to be flexible and adaptable, and as such, the dosing frequency, the doses, and the number of cohorts of BXCL501 allowed for change based on ongoing safety review and medical monitoring of safety, tolerability, and efficacy data after each dose-escalating cohort.

Phase 2 evaluated 6 cohorts (n=25 subjects per cohort according to the 4:1 randomization ratio; n= 20 active BXCL501 and n=5 placebo). The following doses were administered: 30 µg (Cohort 1), 60 µg (Cohort 2), 90 µg (Cohort 3), 120 µg (Cohort 4), and 180 µg (Cohort 5). The dose for Cohort 6 (240 μg) was determined from data acquired from Cohorts 1-5 and Cohort 6 was activated prior to the end of the study.

Other evaluations during the study included establishing the preliminary efficacy of multiple BXCL501 doses relative to placebo and evaluation of pharmacokinetics (PK) in subjects undergoing opiate withdrawal.

ELIGIBILITY:
Inclusion Criteria

1. Male and female subjects who are 18 years of age to less than 65 years of age.
2. Meets criteria for moderate to severe opioid use disorder as per Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria and confirmed by the Mini International Neuropsychiatric Interview (MINI) with physiological dependence as evidenced by a Clinical Opiate Withdrawal (COWS) score of >5 or a positive naloxone challenge upon admission on Day 1.
3. Subjects who can read, understand, and provide written informed consent. Women of childbearing potential must have a negative pregnancy test and agree to be abstinent or use an acceptable method of contraception for the duration of the study.

Exclusion Criteria

1. Positive urine pregnancy test at screening or when tested or currently breast feeding.
2. Clinically significant history of cardiac disease, screening and baseline heart rate of <55 beats per minutes or systolic blood pressure <110 mmHg or diastolic blood pressure <70 mmHg.
3. History or presence of a significant medical disease or disorder which, in the opinion of the investigator, increases the risk or may confound the interpretation of study measures, as confirmed by screening laboratory results.
4. Hepatic dysfunction (marked by ascites, or bilirubin >10% above the upper limit of normal [ULN] or liver function tests >3 x ULN) at the screening visit.
5. Acute active Hepatitis B or C as evidenced by positive serology and aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >2 x ULN.
6. Clinically significant abnormal ECG findings such as second- or third-degree heart block, uncontrolled arrhythmia, or QTcF (Fridericia correction formula) interval >450 msec for males, and >470 msec for females at screening or prior to dosing.
7. Any psychiatric disorder that would compromise ability to complete study requirements.
8. Currently meets DSM-5 criteria for substance abuse disorder, moderate or severe for any substance other than opioids, caffeine, or nicotine and/or current physical dependence on drugs that pose risk of withdrawal that requires medical management such as alcohol or benzodiazepines.
9. History of suicidal behavior within the last 1 year prior to screening.
10. Participation in a clinical trial of a non-FDA-approved pharmacological agent within 30 days prior to screening.
11. Use of any excluded medication at screening or anticipated/required use during the study period.
12. Subjects with a history of intolerance to morphine.
13. Any finding that, in the view of the principal investigator, would compromise the subject's ability to fulfill the protocol visit schedule or visit requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Risinger, MD, Study Director — Chief Medical Officer
Locations (3):
- United States (3):
  - BioXcel Clinical Research Site, Miami Lakes, Florida
  - BioXcel Clinical Research Site, Marlton, New Jersey
  - BioXcel Clinical Research Site, New York, New York

IPD SHARING:
Plan to Share IPD: No
The Study Protocol and Statistical Analysis Plan (SAP) will be shared. Individual data is summarized by treatment group.

REFERENCES:
- [Background] Jones JD, Rajachandran L, Yocca F, Risinger R, De Vivo M, Sabados J, Levin FR, Comer SD. Sublingual dexmedetomidine (BXCL501) reduces opioid withdrawal symptoms: findings from a multi-site, phase 1b/2, randomized, double-blind, placebo-controlled trial. Am J Drug Alcohol Abuse. 2023 Jan 2;49(1):109-122. doi: 10.1080/00952990.2022.2144743. Epub 2023 Jan 11. PMID 36630319

RESULTS

PARTICIPANT FLOW:
Groups:
- Morphine Maintenance, Then Cohort 1- 30 Micrograms: Oral morphine 30 mg immediate tablets, then sublingual film containing 30 micrograms BXCL501 (Dexmedetomidine)
- Morphine Maintenance, Then Cohort 2- 60 Micrograms: Oral morphine 30 mg immediate tablets, then sublingual film containing 60 micrograms BXCL501 (Dexmedetomidine)
- Morphine Maintenance, Then Cohort 3- 90 Micrograms: Oral morphine 30 mg immediate tablets, then sublingual film containing 90 micrograms BXCL501 (Dexmedetomidine)
- Morphine Maintenance, Then Cohort 4- 120 Micrograms: Oral morphine 30 mg immediate tablets, then sublingual film containing 120 micrograms BXCL501 (Dexmedetomidine)
- Morphine Maintenance, Then Cohort 5- 180 Micrograms: Oral morphine 30 mg immediate tablets, then sublingual film containing 180 micrograms BXCL501 (Dexmedetomidine)
- Morphine Maintenance, Then Cohort 6- 240 Micrograms: Oral morphine 30 mg immediate tablets, then sublingual film containing 240 micrograms BXCL501 (Dexmedetomidine)
- Morphine Maintenance, Then Cohort 7- Placebo: Oral morphine 30 mg immediate tablets, then sublingual film containing placebo
Period: Opioid Maintenance Phase
Arm/Group | Morphine Maintenance, Then Cohort 1- 30 Micrograms | Morphine Maintenance, Then Cohort 2- 60 Micrograms | Morphine Maintenance, Then Cohort 3- 90 Micrograms | Morphine Maintenance, Then Cohort 4- 120 Micrograms | Morphine Maintenance, Then Cohort 5- 180 Micrograms | Morphine Maintenance, Then Cohort 6- 240 Micrograms | Morphine Maintenance, Then Cohort 7- Placebo
Started | 29 | 35 | 31 | 32 | 40 | 33 | 25
Completed | 17 | 17 | 21 | 19 | 21 | 15 | 25
Not Completed | 12 | 18 | 10 | 13 | 19 | 18 | 0
Period: Double-blind Treatment Phase
Arm/Group | Morphine Maintenance, Then Cohort 1- 30 Micrograms | Morphine Maintenance, Then Cohort 2- 60 Micrograms | Morphine Maintenance, Then Cohort 3- 90 Micrograms | Morphine Maintenance, Then Cohort 4- 120 Micrograms | Morphine Maintenance, Then Cohort 5- 180 Micrograms | Morphine Maintenance, Then Cohort 6- 240 Micrograms | Morphine Maintenance, Then Cohort 7- Placebo
Started | 17 | 17 | 21 | 19 | 21 | 15 | 25
Completed | 7 | 5 | 6 | 7 | 5 | 6 | 6
Not Completed | 10 | 12 | 15 | 12 | 16 | 9 | 19
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 12 | 15 | 11 | 15 | 9 | 19

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1- 30 Micrograms: Sublingual film containing 30 Micrograms Dexmedetomidine or Placebo
  Dexmedetomidine (BXCL501): Sublingual Film
  Placebo: Sublingual Placebo film
- Cohort 2- 60 Micrograms: Sublingual film containing 60 Micrograms Dexmedetomidine or Placebo
  Dexmedetomidine (BXCL501): Sublingual Film
  Placebo: Sublingual Placebo film
- Cohort 3- 90 Micrograms: Sublingual film containing 90 Micrograms Dexmedetomidine or Placebo
  Dexmedetomidine (BXCL501): Sublingual Film
  Placebo: Sublingual Placebo film
- Cohort 4- 120 Micrograms: Sublingual film containing 120 Micrograms Dexmedetomidine or Placebo
  Dexmedetomidine (BXCL501): Sublingual Film
  Placebo: Sublingual Placebo film
- Cohort 5- 180 Micrograms: Sublingual film containing 180 Micrograms Dexmedetomidine or Placebo
  Dexmedetomidine (BXCL501): Sublingual Film
  Placebo: Sublingual Placebo film
- Cohort 6- 240 Micrograms: Sublingual film containing 240 Micrograms Dexmedetomidine or Placebo
  Dexmedetomidine (BXCL501): Sublingual Film
  Placebo: Sublingual Placebo film
- Pooled Placebo: Placebo: Sublingual Placebo film
- Total: Total of all reporting groups
Arm/Group | Cohort 1- 30 Micrograms | Cohort 2- 60 Micrograms | Cohort 3- 90 Micrograms | Cohort 4- 120 Micrograms | Cohort 5- 180 Micrograms | Cohort 6- 240 Micrograms | Pooled Placebo | Total
Number analyzed (Participants) | 17 | 17 | 21 | 19 | 21 | 15 | 25 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (13.88) | 45.5 (12.56) | 39.3 (9.64) | 41.3 (9.55) | 42.9 (9.57) | 42.0 (11.86) | 42.1 (10.97) | 42.0 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 2 | 4 | 6 | 4 | 6 | 36
  Male | 11 | 9 | 19 | 15 | 15 | 11 | 19 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 5 | 2 | 4 | 4 | 2 | 18
  Not Hispanic or Latino | 16 | 17 | 16 | 17 | 17 | 11 | 23 | 117
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 10 | 4 | 6 | 7 | 5 | 9 | 48
  White | 10 | 7 | 16 | 12 | 13 | 10 | 16 | 84
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Height [Mean (Standard Deviation); unit: cm] | 170.32 (6.933) | 170.14 (7.255) | 176.46 (10.176) | 171.57 (10.942) | 172.25 (10.349) | 174.17 (7.998) | 174.42 (9.220) | 172.92 (9.283)
Weight [Mean (Standard Deviation); unit: kg] | 71.22 (10.604) | 66.38 (10.159) | 78.05 (13.827) | 82.04 (17.999) | 83.65 (26.189) | 83.51 (21.313) | 79.23 (21.480) | 77.98 (19.085)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.65 (4.135) | 22.95 (3.217) | 25.05 (3.824) | 28.16 (7.856) | 28.05 (8.248) | 27.47 (6.589) | 26.21 (7.721) | 26.12 (6.498)

OUTCOME MEASURES:

1. Primary Outcome: Peak SOWS Scores at Baseline and Over Time
Description: Short Opiate Withdrawal Scale (SOWS)-Gossop: The SOWs scale is a validated 10-item patient-reported scale designed to measure the symptoms of withdrawal in subjects who are dependent on opioids. Each of the 10 items represents a symptom: "feeling sick," "stomach cramps," "muscle spasms/twitching," "feeling of coldness," "heart pounding," "muscular tension," "aches and pains," "yawning," "runny eyes," and "insomnia/problems sleeping." Scores on the SOWS-Gossop can range from 0 to 30, with higher scores indicating greater severity of withdrawal symptoms.
Time Frame: Baseline (pre-dose day 6) and at days 6, 7, 8, 9, 10, 11, 12, 13, and 14 post-dose
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 30 Micrograms: Sublingual film containing 30 Micrograms Dexmedetomidine
  Dexmedetomidine (BXCL501): Sublingual Film
- 60 Micrograms: Sublingual film containing 60 Micrograms Dexmedetomidine
  Dexmedetomidine (BXCL501): Sublingual Film
- 90 Micrograms: Sublingual film containing 90 Micrograms Dexmedetomidine
  Dexmedetomidine (BXCL501): Sublingual Film
- 120 Micrograms: Sublingual film containing 120 Micrograms Dexmedetomidine
  Dexmedetomidine (BXCL501): Sublingual Film
- 180 Micrograms: Sublingual film containing 180 Micrograms Dexmedetomidine
  Dexmedetomidine (BXCL501): Sublingual Film
- 240 Micrograms: Sublingual film containing 240 Micrograms Dexmedetomidine
  Dexmedetomidine (BXCL501): Sublingual Film
- Pooled Placebo: Sublingual film containing Placebo
  Comparator: Placebo Sublingual Film
Arm/Group | 30 Micrograms | 60 Micrograms | 90 Micrograms | 120 Micrograms | 180 Micrograms | 240 Micrograms | Pooled Placebo
Number analyzed (Participants) | 17 | 17 | 21 | 19 | 21 | 15 | 24
score on a scale
  Baseline, Pre-Dose, Day 6 | 3.6 (3.24) | 5.2 (3.86) | 6.0 (5.45) | 4.7 (4.64) | 5.0 (4.43) | 6.5 (7.38) | 6.2 (6.93)
  Day 6 Post-dose: number analyzed (Participants) | 17 | 16 | 20 | 19 | 21 | 15 | 24
  Day 6 Post-dose | 4.0 (3.30) | 9.1 (7.49) | 7.7 (5.01) | 8.6 (7.05) | 9.0 (7.20) | 11.2 (6.27) | 7.5 (7.08)
  Day 7 Post-dose: number analyzed (Participants) | 13 | 12 | 18 | 13 | 16 | 12 | 14
  Day 7 Post-dose | 8.8 (8.19) | 9.6 (7.09) | 9.3 (6.10) | 10.7 (7.20) | 14.9 (9.42) | 14.2 (11.17) | 10.2 (8.10)
  Day 8 Post-dose: number analyzed (Participants) | 13 | 7 | 16 | 10 | 16 | 10 | 13
  Day 8 Post-dose | 9.8 (7.86) | 7.4 (7.23) | 8.6 (5.86) | 8.0 (6.46) | 10.8 (7.63) | 12.0 (7.59) | 9.1 (7.50)
  Day 9 Post-dose: number analyzed (Participants) | 9 | 7 | 10 | 10 | 12 | 8 | 8
  Day 9 Post-dose | 6.8 (3.35) | 6.0 (3.27) | 6.5 (4.72) | 6.9 (6.44) | 10.2 (6.44) | 11.5 (9.27) | 8.0 (9.74)
  Day 10 Post-dose: number analyzed (Participants) | 7 | 6 | 7 | 8 | 11 | 6 | 7
  Day 10 Post-dose | 6.7 (6.02) | 4.3 (2.66) | 5.3 (5.28) | 4.6 (5.87) | 8.5 (5.22) | 8.5 (5.32) | 4.1 (3.80)
  Day 11 Post-dose: number analyzed (Participants) | 7 | 5 | 7 | 8 | 11 | 15 | 24
  Day 11 Post-dose | 4.0 (3.96) | 3.8 (4.38) | 3.4 (3.64) | 2.5 (2.56) | 7.2 (6.34) | 4.8 (3.25) | 5.1 (8.57)
  Day 12 Post-dose: number analyzed (Participants) | 7 | 5 | 6 | 8 | 11 | 6 | 6
  Day 12 Post-dose | 5.4 (5.65) | 3.2 (3.03) | 2.8 (3.54) | 2.9 (3.83) | 5.7 (5.10) | 5.2 (3.76) | 7.0 (11.38)
  Day 13 Post-dose: number analyzed (Participants) | 7 | 5 | 6 | 8 | 7 | 6 | 6
  Day 13 Post-dose | 5.0 (4.12) | 5.4 (6.99) | 4.0 (3.90) | 4.0 (4.57) | 3.3 (2.29) | 3.5 (1.38) | 4.3 (6.22)
  Day 14 Post-dose: number analyzed (Participants) | 7 | 5 | 6 | 7 | 6 | 6 | 6
  Day 14 Post-dose | 2.4 (2.64) | 2.8 (3.83) | 2.7 (3.88) | 2.1 (2.54) | 1.7 (2.34) | 1.2 (1.83) | 4.3 (9.67)

2. Secondary Outcome: Peak COWS Score at Baseline and Over Time
Description: Clinical Opiate Withdrawal Scale (COWS): The COWS scale is a validated, 11-item questionnaire designed to quantify withdrawal symptoms. Symptoms evaluated include resting pulse rate, sweating, restlessness, pupil size, bone or joint aches, runny nose or tearing, gastrointestinal upset, tremor, yawning, anxiety or irritability, and gooseflesh. COWS total scores range from 0 to 48, with 5 to 12 indicating mild symptoms, 13 to 24 indicating moderate symptoms, 25 to 36 indicating moderately severe symptoms, and greater than 36 indicating severe symptoms.
Time Frame: Baseline (pre-dose day 6) and at days 6, 7, 8, 9, 10, 11, 12, 13, and 14 post-dose
Population: Full Analysis Set (FAS):
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 30 Micrograms | 60 Micrograms | 90 Micrograms | 120 Micrograms | 180 Micrograms | 240 Micrograms | Pooled Placebo
Number analyzed (Participants) | 17 | 17 | 21 | 19 | 21 | 15 | 24
score on a scale
  Baseline (Pre-Dose, Day 6) | 2.4 (1.77) | 4.6 (3.54) | 5.2 (3.87) | 4.1 (2.68) | 4.4 (3.07) | 3.8 (2.76) | 2.7 (2.49)
  Day 6 Post dose: number analyzed (Participants) | 17 | 16 | 20 | 19 | 21 | 15 | 24
  Day 6 Post dose | 4.2 (2.77) | 6.7 (3.16) | 4.6 (2.28) | 4.1 (2.56) | 5.4 (3.17) | 6.7 (3.83) | 5 (2.83)
  Day 7 Postdose: number analyzed (Participants) | 13 | 12 | 18 | 13 | 16 | 12 | 14
  Day 7 Postdose | 8.8 (5.37) | 6.1 (3.73) | 6.1 (2.32) | 6.5 (3.07) | 7.4 (3.65) | 7.3 (4.29) | 6.1 (3.25)
  Day 8 Postdose: number analyzed (Participants) | 13 | 7 | 16 | 10 | 16 | 10 | 14
  Day 8 Postdose | 8.9 (5.54) | 4.3 (3.4) | 6.1 (3.93) | 4.8 (2.86) | 6.8 (3.64) | 6.0 (4.29) | 5.9 (3.61)
  Day 9 Postdose: number analyzed (Participants) | 9 | 7 | 10 | 10 | 12 | 8 | 9
  Day 9 Postdose | 6.2 (3.80) | 4.7 (1.98) | 4.7 (2.54) | 3.5 (2.22) | 7.0 (3.30) | 6.8 (3.01) | 6.0 (6.14)
  Day 10 Postdose: number analyzed (Participants) | 7 | 6 | 7 | 10 | 11 | 6 | 8
  Day 10 Postdose | 4.9 (3.67) | 3.5 (1.52) | 3.7 (2.56) | 3.5 (2.07) | 4.6 (1.91) | 3.8 (1.47) | 3.9 (2.17)
  Day 11 Postdose: number analyzed (Participants) | 7 | 5 | 7 | 8 | 11 | 6 | 7
  Day 11 Postdose | 5.4 (4.28) | 5.0 (5.83) | 2.0 (1.63) | 3.4 (2.20) | 4.5 (3.33) | 3.5 (2.26) | 3.0 (2.83)
  Day 12 Postdose: number analyzed (Participants) | 7 | 5 | 6 | 8 | 11 | 6 | 6
  Day 12 Postdose | 3.6 (2.07) | 4.6 (4.28) | 2.0 (1.10) | 2.4 (1.77) | 3.6 (2.46) | 3.3 (1.75) | 4.5 (4.76)
  Day 13 Postdose: number analyzed (Participants) | 7 | 5 | 6 | 8 | 7 | 6 | 6
  Day 13 Postdose | 5.3 (2.93) | 4.0 (3.67) | 4.2 (2.93) | 2.5 (1.77) | 2.6 (1.27) | 3.0 (2.10) | 3.2 (3.97)
  Day 14 Postdose: number analyzed (Participants) | 7 | 5 | 6 | 7 | 6 | 6 | 6
  Day 14 Postdose | 3.4 (1.99) | 3.2 (2.17) | 2.8 (2.32) | 1.4 (1.62) | 2.3 (1.37) | 3.3 (2.42) | 3.5 (3.56)

3. Secondary Outcome: Average COWS Scores at Baseline and Over Time
Description: as for outcome 2
Time Frame: Baseline (pre-dose day 6) and at days 6, 7, 8, 9, 10, 11, 12, 13, and 14 post-dose
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 30 Micrograms | 60 Micrograms | 90 Micrograms | 120 Micrograms | 180 Micrograms | 240 Micrograms | Pooled Placebo
Number analyzed (Participants) | 17 | 17 | 21 | 19 | 21 | 15 | 24
score on a scale
  Baseline (Pre-Dose, Day 6): number analyzed (Participants) | 17 | 16 | 20 | 19 | 21 | 15 | 24
  Baseline (Pre-Dose, Day 6) | 2.41 (1.770) | 4.59 (3.537) | 5.19 (3.868) | 4.05 (2.677) | 4.38 (3.074) | 3.80 (2.757) | 2.71 (2.493)
  Day 6, Post-Dose | 3.21 (1.913) | 5.22 (3.173) | 3.85 (2.254) | 3.26 (2.287) | 4.29 (2.853) | 4.83 (2.814) | 4.02 (2.477)
  Day 7 Post dose: number analyzed (Participants) | 13 | 12 | 18 | 13 | 16 | 12 | 14
  Day 7 Post dose | 6.19 (4.013) | 5.63 (3.562) | 4.92 (2.390) | 5.08 (2.849) | 6.41 (3.205) | 6.04 (4.109) | 4.54 (2.349)
  Day 8 Post dose: number analyzed (Participants) | 13 | 7 | 16 | 10 | 16 | 10 | 14
  Day 8 Post dose | 7.19 (4.489) | 3.21 (2.797) | 5.19 (3.646) | 3.70 (2.163) | 5.81 (3.391) | 4.40 (2.569) | 5.14 (3.359)
  Day 9 Post dose: number analyzed (Participants) | 9 | 7 | 10 | 10 | 12 | 8 | 9
  Day 9 Post dose | 5.11 (3.462) | 3.50 (1.780) | 4.20 (2.440) | 2.80 (1.859) | 5.63 (2.970) | 5.25 (2.478) | 5.39 (6.279)
  Day 10 Post dose: number analyzed (Participants) | 7 | 6 | 7 | 10 | 11 | 6 | 8
  Day 10 Post dose | 3.43 (2.992) | 3.17 (1.693) | 3.07 (2.110) | 2.70 (1.884) | 3.82 (1.647) | 2.67 (1.252) | 2.81 (1.731)
  Day 11 Postdose: number analyzed (Participants) | 7 | 5 | 7 | 8 | 11 | 6 | 7
  Day 11 Postdose | 3.57 (2.589) | 3.30 (3.054) | 1.50 (1.258) | 2.69 (2.086) | 3.59 (2.782) | 2.58 (1.530) | 2.50 (2.799)
  Day 12 Post dose: number analyzed (Participants) | 7 | 5 | 6 | 8 | 11 | 6 | 6
  Day 12 Post dose | 3.07 (2.263) | 3.30 (2.864) | 1.42 (1.068) | 1.81 (1.438) | 3.14 (2.521) | 2.58 (1.715) | 3.58 (4.364)
  Day 13 Post dose: number analyzed (Participants) | 7 | 5 | 6 | 8 | 7 | 6 | 6
  Day 13 Post dose | 4.07 (2.335) | 3.20 (3.883) | 2.58 (1.594) | 2.13 (1.847) | 1.71 (1.035) | 2.50 (1.549) | 2.58 (3.247)
  Day 14 Post dose: number analyzed (Participants) | 7 | 5 | 6 | 7 | 6 | 6 | 6
  Day 14 Post dose | 3.43 (1.988) | 2.70 (1.924) | 1.92 (1.201) | 1.21 (1.468) | 2.33 (1.366) | 3.00 (1.897) | 3.33 (3.204)

4. Secondary Outcome: Average SOWS at Baseline and Over Time
Description: Short Opiate Withdrawal Scale (SOWS)-Gossop: The SOWs scale is a validated 10-item patient-reported scale designed to measure the symptoms of withdrawal in subjects who are dependent on opioids.5 Each of the 10 items represents a symptom: "feeling sick," "stomach cramps," "muscle spasms/twitching," "feeling of coldness," "heart pounding," "muscular tension," "aches and pains," "yawning," "runny eyes," and "insomnia/problems sleeping." Scores on the SOWS-Gossop can range from 0 to 30, with higher scores indicating greater severity of withdrawal symptoms.
Time Frame: Baseline (pre-dose day 6) and at days 6, 7, 8, 9, 10, 11, 12, 13, and 14 post-dose
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 30 Micrograms | 60 Micrograms | 90 Micrograms | 120 Micrograms | 180 Micrograms | 240 Micrograms | Pooled Placebo
Number analyzed (Participants) | 17 | 17 | 21 | 19 | 21 | 15 | 24
score on a scale
  Baseline, Pre-Dose, Day 6 | 3.59 (3.242) | 5.18 (3.861) | 5.95 (5.454) | 4.74 (4.641) | 4.95 (4.433) | 6.53 (7.376) | 6.21 (6.934)
  Day 6 Postdose: number analyzed (Participants) | 17 | 16 | 20 | 19 | 21 | 15 | 24
  Day 6 Postdose | 3.35 (3.071) | 7.13 (6.617) | 5.88 (3.916) | 5.79 (4.388) | 6.81 (5.815) | 8.50 (4.935) | 6.58 (6.780)
  Day 7 Postdose: number analyzed (Participants) | 13 | 12 | 18 | 13 | 16 | 12 | 14
  Day 7 Postdose | 6.73 (5.426) | 8.83 (6.959) | 7.39 (4.513) | 8.42 (6.380) | 11.53 (7.702) | 10.63 (9.670) | 7.54 (5.458)
  Day 8 Postdose: number analyzed (Participants) | 13 | 7 | 16 | 10 | 16 | 10 | 13
  Day 8 Postdose | 8.65 (7.967) | 4.86 (4.616) | 7.63 (5.614) | 6.85 (5.991) | 9.31 (7.765) | 10.15 (8.267) | 7.92 (6.828)
  Day 9 Postdose: number analyzed (Participants) | 9 | 7 | 10 | 10 | 12 | 8 | 8
  Day 9 Postdose | 6.11 (3.361) | 4.14 (2.428) | 5.65 (4.404) | 4.95 (5.325) | 8.21 (4.398) | 9.00 (7.521) | 7.06 (9.318)
  Day 10 Postdose: number analyzed (Participants) | 7 | 6 | 7 | 10 | 11 | 6 | 8
  Day 10 Postdose | 4.79 (4.030) | 3.33 (2.206) | 4.57 (4.457) | 3.50 (5.217) | 6.59 (3.740) | 5.08 (2.178) | 3.06 (3.076)
  Day 11 Postdose: number analyzed (Participants) | 7 | 5 | 7 | 8 | 11 | 6 | 7
  Day 11 Postdose | 2.79 (2.464) | 2.20 (2.414) | 3.00 (3.651) | 1.94 (2.195) | 5.18 (5.139) | 3.42 (2.223) | 3.50 (6.110)
  Day 12 Postdose: number analyzed (Participants) | 7 | 5 | 6 | 8 | 11 | 6 | 6
  Day 12 Postdose | 4.00 (4.252) | 2.20 (2.168) | 2.00 (2.387) | 2.19 (3.294) | 4.77 (4.967) | 3.67 (2.696) | 4.58 (6.953)
  Day 13 Postdose: number analyzed (Participants) | 7 | 5 | 6 | 8 | 7 | 6 | 6
  Day 13 Postdose | 3.93 (2.775) | 4.70 (7.068) | 2.08 (1.882) | 3.31 (3.891) | 2.21 (1.542) | 2.50 (1.049) | 3.25 (5.760)
  Day 14 Postdose: number analyzed (Participants) | 7 | 5 | 6 | 7 | 6 | 6 | 6
  Day 14 Postdose | 2.43 (2.637) | 2.40 (3.362) | 1.67 (2.251) | 1.71 (2.270) | 1.67 (2.338) | 1.08 (1.686) | 2.92 (6.216)

5. Secondary Outcome: Time to Drop-out After Discontinuation of Opioid Maintenance Phase
Description: Time to drop-out during double-blind treatment phase after discontinuation of opioid maintenance Phase.
Time Frame: Day 6 through Day 14
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | 30 Micrograms | 60 Micrograms | 90 Micrograms | 120 Micrograms | 180 Micrograms | 240 Micrograms | Pooled Placebo
Number analyzed (Participants) | 17 | 17 | 21 | 19 | 21 | 15 | 25
Days | 3.1 [0.7 to NA] — The upper limit is not estimable due to the limitations imposed by the small sample size | 1.5 [0.00 to NA] — The upper limit is not estimable due to the limitations imposed by the small sample size | 3.1 [2.2 to 6.0] | 5.1 [1.1 to NA] — The upper limit is not estimable due to the limitations imposed by the small sample size | 6.1 [2.1 to NA] — The upper limit is not estimable due to the limitations imposed by the small sample size | 3.5 [1.0 to NA] — The upper limit is not estimable due to the limitations imposed by the small sample size | 2.0 [0.7 to 5.1]

6. Secondary Outcome: Number and Percentage of Subject Drop-out After Discontinuation of Opioid Maintenance Phase Maintenance Within Each Treatment Group
Description: Number and Percentage of Subject Drop-out after Discontinuation of Opioid Maintenance Phase Within Each Treatment Group Between Days 6-14.
Time Frame: Day 6 through Day 14
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | 30 Micrograms | 60 Micrograms | 90 Micrograms | 120 Micrograms | 180 Micrograms | 240 Micrograms | Pooled Placebo
Number analyzed (Participants) | 17 | 17 | 21 | 19 | 21 | 15 | 25
Participants
  Day 6 | 3 | 4 | 3 | 3 | 3 | 2 | 7
  Day 7 | 1 | 5 | 2 | 5 | 2 | 4 | 4
  Day 8 | 3 | 0 | 4 | 1 | 4 | 1 | 4
  Day 9 | 3 | 0 | 5 | 0 | 1 | 1 | 2
  Day 10 | 0 | 2 | 0 | 0 | 0 | 1 | 0
  Day 11 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Day 12 | 0 | 0 | 1 | 0 | 2 | 0 | 0
  Day 13 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  Day 14 | 0 | 0 | 0 | 0 | 1 | 0 | 0

7. Secondary Outcome: Total ACES Total Score Over Time - 2 hr. Post-First Dose
Description: Overall Agitation-Calmness Evaluation Scale (ACES): The ACES scale is a single-item measure rating overall agitation and sedation, ranging from 1 (marked agitation) to 9 (unarousable). This outcome measures the total ACES total score over time at 2 hours, post-first dose.
Time Frame: Post-Dose Day 6 to Day 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 30 Micrograms | 60 Micrograms | 90 Micrograms | 120 Micrograms | 180 Micrograms | 240 Micrograms | Pooled Placebo
Number analyzed (Participants) | 17 | 16 | 20 | 19 | 21 | 15 | 25
units on a scale
  Day 6, Post-Dose | 4.6 (1.27) | 3.4 (1.71) | 4.4 (1.35) | 4.9 (1.31) | 4.7 (1.35) | 4.9 (1.73) | 4.3 (1.40)
  Day 7, Post-Dose: number analyzed (Participants) | 13 | 12 | 18 | 13 | 16 | 12 | 14
  Day 7, Post-Dose | 4.3 (0.95) | 3.6 (1.83) | 3.8 (1.29) | 3.9 (0.76) | 4.1 (1.48) | 4.4 (1.73) | 4.1 (0.86)
  Day 8, Post-Dose: number analyzed (Participants) | 13 | 7 | 16 | 11 | 16 | 10 | 14
  Day 8, Post-Dose | 3.8 (1.17) | 4.1 (1.07) | 4.0 (1.26) | 4.6 (1.43) | 4.2 (1.17) | 5.0 (1.83) | 4.1 (0.83)
  Day 9, Post-Dose: number analyzed (Participants) | 9 | 7 | 10 | 10 | 12 | 7 | 8
  Day 9, Post-Dose | 3.0 (0.87) | 4.1 (1.46) | 3.7 (0.67) | 4.5 (1.18) | 3.5 (0.80) | 4.7 (2.06) | 3.8 (0.46)
  Day 10, Post-Dose: number analyzed (Participants) | 7 | 6 | 7 | 10 | 11 | 6 | 8
  Day 10, Post-Dose | 4.1 (1.77) | 3.8 (0.98) | 4.1 (0.38) | 4.3 (1.06) | 4.3 (1.01) | 4.3 (1.37) | 4.4 (0.92)
  Day 11, Post-Dose: number analyzed (Participants) | 7 | 5 | 7 | 8 | 11 | 6 | 7
  Day 11, Post-Dose | 4.7 (1.50) | 4.0 (0.71) | 4.1 (0.38) | 4.1 (0.64) | 3.9 (0.94) | 4.2 (0.41) | 4.6 (1.13)
  Day 12, Post-Dose: number analyzed (Participants) | 7 | 5 | 6 | 8 | 11 | 6 | 6
  Day 12, Post-Dose | 4.3 (0.76) | 4.4 (1.4) | 4.7 (1.21) | 4.0 (0.00) | 4.1 (0.83) | 4.8 (1.33) | 4.0 (1.10)

ADVERSE EVENTS:
Time Frame: 9 days
Description: The number of subjects that experienced at least one Treatment Emergent Adverse Event (TEAE) during the double-blind randomized Phase. Treatment-Emergent Adverse Events (TEAEs) were exclusively documented during the double-blind Phase, aiming to evaluate the safety profile of BXCL501 in the context of opioid withdrawal subsequent to the cessation of oral morphine.
Groups:
- 240 Micrograms: Sublingual film containing 180 Micrograms Dexmedetomidine
  Dexmedetomidine (BXCL501): Sublingual Film
- Pooled Placebo: Sublingual film containing Placebo
  Placebo: Sublingual Placebo film
Arm/Group | 30 Micrograms | 60 Micrograms | 90 Micrograms | 120 Micrograms | 180 Micrograms | 240 Micrograms | Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/21 | 0/19 | 0/21 | 0/15 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/21 | 0/19 | 0/21 | 0/15 | 0/25
Other Adverse Events (participants affected / at risk) | 1/17 | 5/17 | 2/21 | 4/19 | 8/21 | 9/15 | 5/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 Micrograms (N=17) | 60 Micrograms (N=17) | 90 Micrograms (N=21) | 120 Micrograms (N=19) | 180 Micrograms (N=21) | 240 Micrograms (N=15) | Pooled Placebo (N=25)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation Increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furnucle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT04470050/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT04470050/SAP_001.pdf